CLINICAL TRIAL: NCT01040260
Title: Low-Cost Contingency Management for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17RT-0081
Record Dates: First submitted 2009-12-27; First posted 2009-12-29 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Tobacco Use Cessation
Keywords: tobacco use disorder
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder | interventions — Counseling; Tobacco Use Cessation Devices; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingency management (Experimental): Use of tangible rewards for verified abstinence
  Interventions: Behavioral: Contingency management
- Counseling plus nicotine patches (Active Comparator): Counseling plus nicotine patches
  Interventions: Other: Counseling; Drug: Nicotine patches

INTERVENTIONS:
Other: Counseling — Smoking cessation counseling
  Other Names: Smoking cessation counseling
  Arms: Counseling plus nicotine patches
Behavioral: Contingency management — Use of tangible rewards for abstinence from smoking
  Other Names: Low-cost contingency management
  Arms: Contingency management
Drug: Nicotine patches — Nicotine patches
  Other Names: Nicotine replacement
  Arms: Counseling plus nicotine patches

SUMMARY:
An innovative low-cost form of contingency management has been developed in which participants receive the chance to draw vouchers from a fish bowl depending on whether or not their abstinence from tobacco is confirmed by expired-air carbon monoxide. The vouchers can be redeemed for prizes of varying value. This form of contingency management has been shown to be effective in the treatment of a variety of substance use disorders, but has not been investigated in a clinical trial focusing on smoking cessation. Thus, the primary purpose of the proposed study will be to investigate the effects of a low-cost prize-based form of contingency management in the treatment of nicotine dependence. To accomplish this objective, we enrolled 103 current smokers into the study. The participants in Study Arm 1 received the contingency management intervention for 8 weeks, and the participants in Study Arm 2 had their smoking status assessed but did not receive the contingency management intervention. Both interventions received brief counseling and nicotine replacement therapy. The counseling was conducted in two 60-minute individual sessions scheduled one week apart with two follow-up phone calls at weeks 3, 4, and 6.

The primary outcome for this study was biochemically-validated smoking status at 3 months (end of treatment), and at 6- and 12-month follow-up. Both continuous and point-prevalent abstinence rates were determined. Saliva cotinine levels were measured in all participants reporting abstinence at each assessment. This study had 80% power to detect a 10% absolute difference in smoking cessation rates between the two treatment conditions (i.e., a 28% quit rate in Study Arm 1 versus a 18% quit rate in Study Arm 2) with alpha set at 0.05. These estimates included an anticipated 15% loss to follow-up over the 12-month study period.

DETAILED DESCRIPTION:
Contingency management as a treatment for substance use disorders involves the use of tangible rewards for confirmed abstinence. There is preliminary evidence that contingency management shows promise as a smoking cessation intervention. An innovative low-cost form of contingency management has been developed in which participants receive the chance to draw vouchers from a fish bowl depending on whether or not their abstinence from tobacco is confirmed by expired-air carbon monoxide. The vouchers can be redeemed for prizes of varying value. This form of contingency management has been shown to be effective in the treatment of a variety of substance use disorders, but has not been investigated in a clinical trial focusing on smoking cessation. Thus, the primary purpose of the proposed study was to investigate the effects of a low-cost prize-based form of contingency management in the treatment of nicotine dependence. To accomplish this objective, we enrolled 103 current smokers into the study. The participants in Study Arm 1 received the contingency management intervention for 8 weeks, and the participants in Study Arm 2 had their smoking status assessed but did not receive the contingency management intervention. Both interventions received brief counseling and nicotine replacement therapy. The counseling was conducted in two 60-minute individual sessions scheduled one week apart with two follow-up phone calls at weeks 3, 4, and 6.

The primary outcome for this study was biochemically-validated smoking status at 3 months (end of treatment), and at 6- and 12-month follow-up. Both continuous and point-prevalent abstinence rates were determined. Saliva cotinine levels were measured in all participants reporting abstinence at each assessment. This study had 80% power to detect a 10% absolute difference in smoking cessation rates between the two treatment conditions (i.e., a 28% quit rate in Study Arm 1 versus a 18% quit rate in Study Arm 2) with alpha set at 0.05. These estimates included an anticipated 15% loss to follow-up over the 12-month study period.

ELIGIBILITY:
Inclusion Criteria:

* Smoke at least 5 cigarettes per day
* Interested in quitting

Exclusion Criteria:

* Cognitive impairment or unstable psychotic disorder that would significantly interfere with the individual's ability to participate in the study.
* Self-reported problem with alcohol or other drugs during the past three months
* Current use of any smoking cessation medication
* Presence of any contraindications for nicotine patches, lozenges, or gum
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Carmody, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- VA Medical Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Counseling Plus Nicotine Patches: Counseling plus nicotine patches, carbon monoxide (CO) testing without contingency management
Period: Overall Study
Arm/Group | Contingency Management | Counseling Plus Nicotine Patches
Started | 53 | 50
Completed | 38 | 39
Not Completed | 15 | 11
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Counseling Plus Nicotine Patches: Counseling plus nicotine patches, CO testing without contingency management
- Total: Total of all reporting groups
Arm/Group | Contingency Management | Counseling Plus Nicotine Patches | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 49 | 100
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (13.5) | 47.3 (12.0) | 46.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 41 | 39 | 80
Region of Enrollment [Number; unit: participants]
  United States | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: Abstinence Rate
Description: Number of participants who abstained from smoking during the 7 day period verified by CO testing
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | Contingency Management | Counseling Plus Nicotine Patches
Number analyzed (Participants) | 53 | 50
participants | 8 | 10

ADVERSE EVENTS:
Time Frame: Participants are asked about adverse at each follow-up assessment visit.
Arm/Group | Contingency Management | Counseling Plus Nicotine Patches
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/50
Other Adverse Events (participants affected / at risk) | 2/53 | 2/50
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contingency Management (N=53) | Counseling Plus Nicotine Patches (N=50)
skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes